CLINICAL TRIAL: NCT02422407
Title: A Biomarker Study to Determine the Gene Expression Signatures of Salivary Gland and Blood in Subjects With Incident Primary Sjögren's Syndrome, Subjects With Sicca, and Healthy Volunteers
Brief Title: A Longitudinal, Observational Biomarker Study in Participants With Primary Sjogren's Syndrome
Status: Completed | Type: Observational
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Other Study IDs: 999SJ001
Record Dates: First submitted 2015-03-19; First posted 2015-04-21 (Estimated); Last update posted 2018-01-19 (Actual); Status verified 2018-01

CONDITIONS: Healthy; Sicca Syndrome; Sjögren's Syndrome
MeSH Terms: conditions — Sjogren's Syndrome | interventions — Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A lip biopsy is taken to determine Sjogrens diagnosis.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Subgroup 1: Healthy Volunteers - subset of which 10 will receive salivary gland biopsy.
  Interventions: Procedure: Biopsy
- Subgroup 2: Diagnosis of pSS based on the criteria of the American-European Consensus Criteria for Sjögren's Syndrome (AECCSS) with positive biopsy result.
  Interventions: Procedure: Biopsy
- Subgroup 3: Diagnosis of pSS based on the criteria of the American-European Consensus Criteria for Sjögren's Syndrome (AECCSS) with negative biopsy result.
  Interventions: Procedure: Biopsy
- Subgroup 4: Presenting with sicca but not satisfying the criteria of the AECCSS for diagnosis of pSS.
  Interventions: Procedure: Biopsy

INTERVENTIONS:
Procedure: Biopsy — Salivary Gland

SUMMARY:
The main objective of the study is to characterize the gene expression in immune and epithelial cells in salivary gland biopsy samples and blood of pSS (primary Sjögren's syndrome) and non-pSS participants including healthy volunteers.

ELIGIBILITY:
Key Inclusion Criteria:

For Healthy Volunteers:

* In good overall health as determined by the Investigator For Participants With Sicca
* Subjects should present with sicca (i.e., dry eyes and dry mouth) at Baseline
* Must be willing to undergo a minor salivary gland (labial) biopsy

Key Exclusion Criteria:

* A history of any clinically significant medical condition, as determined by the Investigator, that may impact study analyses
* A chronic or persistent infection human immunodeficiency virus (HIV), hepatitis B, hepatitis C, and/or tuberculosis
* Pre-existing connective tissue disease or autoimmune disease, such as systemic lupus erythematosus (SLE), rheumatoid arthritis, systemic sclerosis, or sarcoidosis
* Any known contraindications of sialoscintigraphy

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants with sicca and healthy volunteers will be recruited from multiple sites
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2015-03-26 (Actual); Primary Completion 2017-08-22 (Actual); Study Completion 2017-08-22 (Actual)

PRIMARY OUTCOMES:
Gene expression levels in immune cells (innate and adaptive) in salivary gland biopsy samples from participants with and without pSS including healthy volunteers | Up to 12 months
Gene expression levels in immune cells (innate and adaptive) in blood samples from participants with and without pSS including healthy volunteers | Up to 12 months
Gene expression levels in epithelial cells in salivary gland biopsy samples from participants with and without pSS including healthy volunteers | Up to 12 months
Gene expression levels in epithelial cells in blood samples from participants with and without pSS including healthy volunteers | Up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (4):
- United States (4):
  - Research Site, Hartford, Connecticut
  - Research Site, Boston, Massachusetts
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Dallas, Texas